CLINICAL TRIAL: NCT01976728
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study Evaluating Three Doses of Subcutaneous Pulsatile GnRH Administered Via OmniPod Pump for Ovulation Induction in Female Subjects With Primary Amenorrhea With Hypogonadotropic Hypogonadism
Brief Title: LutrePulse Hypogonadotropic Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000070
Record Dates: First submitted 2013-10-15; First posted 2013-11-06 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-01

CONDITIONS: Primary Amenorrhea With Hypogonadotropic Hypogonadism
MeSH Terms: interventions — Pulse; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- LutrePulse 10 µg/pulse (Experimental): Gonadorelin acetate 10 µg/pulse
  Interventions: Drug: Gonadorelin acetate subcutaneous (SC) 10 μg/pulse as a fixed dose, administered via. OmniPod pump
- LutrePulse 15 µg/pulse (Experimental): Gonadorelin acetate 15 µg/pulse
  Interventions: Drug: Gonadorelin acetate SC 15 μg/pulse as a fixed dose, administered via. OmniPod pump
- LutrePulse 20 µg/pulse (Experimental): Gonadorelin acetate 20 µg/pulse
  Interventions: Drug: Gonadorelin acetate SC 20 μg/pulse as a fixed dose, administered via. OmniPod pump
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo (SC 10, 15, or 20 μg/pulse as a fixed dose, administered via. OmniPod pump)

INTERVENTIONS:
Drug: Gonadorelin acetate subcutaneous (SC) 10 μg/pulse as a fixed dose, administered via. OmniPod pump
  Other Names: LutrePulse
  Arms: LutrePulse 10 µg/pulse
Drug: Gonadorelin acetate SC 15 μg/pulse as a fixed dose, administered via. OmniPod pump
  Other Names: LutrePulse
  Arms: LutrePulse 15 µg/pulse
Drug: Gonadorelin acetate SC 20 μg/pulse as a fixed dose, administered via. OmniPod pump
  Other Names: LutrePulse
  Arms: LutrePulse 20 µg/pulse
Drug: Placebo (SC 10, 15, or 20 μg/pulse as a fixed dose, administered via. OmniPod pump)
  Arms: Placebo

SUMMARY:
To compare the ovulation rate in women with primary amenorrhea with hypogonadotropic hypogonadism following pulsatile gonadotropin-releasing hormone (GnRH) treatment using the OmniPod pump versus placebo

ELIGIBILITY:
Inclusion Criteria:

* Women 18-40 years old
* Body mass index (BMI) between 18 and 38 kg/m2
* Clinical history or recently diagnosed with primary amenorrhea with hypogonadotropic hypogonadism
* Hormonal values in a centrally analyzed fasting blood sample: FSH <5 IU/L and mean LH <5 IU/L
* Desire to become pregnant
* Discontinued estrogen-progesterone replacement therapy at least 1 month before screening
* Negative progestin challenge test performed during screening
* PAP smear within 24 months of the initial visit
* Normal or stable CT scan or MRI scan of the hypothalamic pituitary region
* Prolactin and thyroid-stimulating hormone (TSH) within normal clinical laboratory limits
* Male partner with normal semen analysis, including volume, liquefaction time, sperm count, and motility, according to the local laboratory normal criteria, within the past year
* Normal transvaginal ultrasound at screening with respect to uterus and adnexa (presence of both ovaries and tubes, without evidence of clinically significant abnormality) and with normal uterine cavity and normal cervix
* Tube patency on saline tubal perfusion, hysterosalpingography or laparoscopy on file within the past 2 years

Exclusion Criteria:

* Any medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the drug
* A history of, or currently diagnosed with clinically important cardiovascular, pulmonary (e.g. serious corticosteroid-dependent asthma), gastrointestinal, hepatic, metabolic, renal, endocrinological (e.g. insulin dependent diabetes mellitus), or neurological (e.g. epilepsy, serious migraine, central nervous system (CNS) lesions (in cases where hypogonadotropic hypogonadism is secondary to a CNS lesion or its treatment) abnormality
* A history of adrenal or uncontrolled thyroid disorders, or hyperprolactinemia
* Prior treatment cycle with gonadotropins or GnRH within the last 2 months
* Known allergy to study drug or its components
* Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Ovarian enlargement or cyst of unknown etiology
* Abnormal gynecological bleeding of undetermined origin
* Previous or current hormone-dependent tumor
* Known active substance abuse
* Planning to undergo in vitro fertilization procedure in the course of a study treatment cycle
* Currently undergoing treatment with gonadotropin hormones (FSH and LH), psychotropic medication, sex hormones, or any other medication known to interfere with normal reproductive function or that can affect GnRH secretion (e.g. neuroleptics, dopamine antagonists, spironolactone, levodopa, phenothiazine, digoxin)
* Ongoing pregnancy or lactation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (35):
- United States (33):
  - Fertility Treatment Center, Tempe, Arizona
  - Center for Reproductive Health UCSF, San Francisco, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - Reproductive Associates of Delaware, Newark, Delaware
  - Columbia Fertility Associates, Washington D.C., District of Columbia
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Center for Reproductive Medicine, Orlando, Florida
  - Georgia Reproductive Specialists, Atlanta, Georgia
  - Fertility Centers of Illinois, Chicago, Illinois
  - Cypress Medical Research Center, Wichita, Kansas
  - Bluegrass Clinical Research Inc., Louisville, Kentucky
  - Maine Medical Center-REI, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State University Physicians Group, Southfield, Michigan
  - Weill Cornell Medical College, New York, New York
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Institute for Reproductive Health, Cincinnati, Ohio
  - University of Cincinnati Physicians, Cincinnati, Ohio
  - UH Case Medical Center, MacDonald Clinical Trials, Cleveland, Ohio
  - Ohio Reproductive Medicine, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Abington IVF & Genetics, L.P., Oklahoma City, Oklahoma
  - Abington Reproductive Medicine, PC, Abington, Pennsylvania
  - Main Line Fertility Center, Bryn Mawr, Pennsylvania
  - Penn State MS Hershey Medical Center, Penn State College of Medicine, Hershey, Pennsylvania
  - University of Pittsburgh, Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Fertility Associates of Memphis PLLC, Memphis, Tennessee
  - Center for Assisted Reproduction, Bedford, Texas
  - Houston Fertility Institute, Houston, Texas
  - Center of Reproductive Medicine, Webster, Texas
  - Utah Fertility Center, Pleasant Grove, Utah
  - Jones Institute for Reproductive Medicine, Norfolk, Virginia
- Canada (2):
  - Olive Fertility Centre, Vancouver, British Columbia
  - Ovo, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 sites randomized subjects to the trial between April 2014 and February 2018. The trial sites that randomized subjects to the trial were: 22 in the United States of America and 2 in Canada.
Pre-assignment Details: A total of 54 subjects were screened, of which 39 subjects were randomized. Of the 39 randomized subjects, 10 were randomized to LutrePulse 10 μg/pulse, 9 were randomized to LutrePulse 15 μg/pulse, 10 were randomized to LutrePulse 20 μg/pulse and 10 were randomized to placebo.
Groups:
- LutrePulse 10 µg/Pulse: Gonadorelin acetate subcutaneous (SC) 10 μg/pulse as a fixed dose, administered via. OmniPod pump
- LutrePulse 15 µg/Pulse: Gonadorelin acetate SC 15 μg/pulse as a fixed dose, administered via. OmniPod pump
- LutrePulse 20 µg/Pulse: Gonadorelin acetate SC 20 μg/pulse as a fixed dose, administered via. OmniPod pump
- Placebo: Placebo (SC 10, 15, or 20 μg/pulse as a fixed dose, administered via. OmniPod pump)
Period: Overall Study
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Started | 10 | 9 | 10 | 10
Dosed | 10 | 9 | 10 | 10
Completed | 9 | 9 | 10 | 10
Not Completed | 1 | 0 | 0 | 0
Not completed — Subject missed multiple doses of IMP | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set comprised all randomized subjects.
Groups:
- LutrePulse 10 µg/Pulse: Gonadorelin acetate SC 10 μg/pulse as a fixed dose, administered via. OmniPod pump
- Total: Total of all reporting groups
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 10 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (4.20) | 29.6 (6.02) | 30.9 (5.67) | 29.5 (2.55) | 30.2 (4.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 10 | 10 | 39
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 3 | 9
  Not Hispanic or Latino | 7 | 7 | 9 | 7 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 0 | 4
  White | 9 | 7 | 7 | 8 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.41 (6.065) | 23.70 (4.567) | 26.53 (4.218) | 23.85 (3.953) | 25.93 (5.159)

OUTCOME MEASURES:

1. Primary Outcome: Ovulation Rate
Description: Calculated as a proportion of subjects with at least 1 post-baseline progesterone level ≥ 6 ng/mL or subjects with confirmed positive serum β-human chorionic gonadotropin (β-hCG) (i.e., 2 positive results) or subjects with a gestational sac documented by transvaginal ultrasound (TVUS).
Time Frame: From treatment Day 1 up to 4 weeks after second positive β-hCG test, approximately 9 weeks
Population: The full analysis set (FAS) comprised all randomized subjects who were included in ITT analysis set and had received at least 14 days of investigational medicinal product (IMP). One subject in the LutrePulse 10 µg/Pulse group was discontinued from the trial after 6 days exposure and is not included in the FAS (LutrePulse 10 µg/Pulse: n=9).
Measure: Count of Participants; unit: Participants
Groups:
- Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled: Gonadorelin acetate SC 15 μg/pulse and SC 20 μg/pulse, administered via. OmniPod pump pooled
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 18 | 10
Participants | 1 | 4 | 5 | 9 | 0
Statistical Analysis 1: Comparison: Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled vs Placebo; The primary efficacy analysis compared the pooled ovulation rate of the LutrePulse 15 μg and 20 μg group to placebo; Test type: Superiority — The hypotheses were tested using a stratified one-sided Fisher's exact test in the FAS including the randomization scheme as the stratification factor; p = 0.0120, Fisher Exact — The SAS PROC FREQ with permutation-based Cochran-Mantel-Haenszel test with exact p-value derived from all possible permutations was employed for the calculation of p-value for the stratified Fisher's exact test; The success threshold at each analysis corresponded to a nominal p-value <0.0130 to maintain an overall one-sided type I error rate of 0.025

2. Secondary Outcome: Progesterone (P4) Levels
Description: Proportion of participants with at least 1 post-baseline P4 level ≥ 10 ng/mL.
Time Frame: Treatment Days 19, 21, 23, 25, and 27
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- LutrePulse 10 µg/Pulse: Gonadorelin acetate SC 10 µg/pulse as a fixed dose, administered via. OmniPod pump
- LutrePulse 15 µg/Pulse: Gonadorelin acetate SC 15 µg/pulse as a fixed dose, administered via. OmniPod pump
- LutrePulse 20 µg/Pulse: Gonadorelin acetate SC 20 µg/pulse as a fixed dose, administered via. OmniPod pump
- Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled: Gonadorelin acetate SC 15 μg/pulse and 20 μg/pulse, administered via. OmniPod pump pooled
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 19 | 10
Participants | 1 | 4 | 3 | 7 | 0
Statistical Analysis 1: Comparison: Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled vs Placebo; P4 levels of the pooled LutrePulse 15 μg and 20 μg group were compared to placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0553, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Clinical Pregnancy Rate
Description: Proportion of subjects with presence of gestational sac and fetal heart movement on TVUS after a second positive serum β-hCG test.
Time Frame: 2 to 4 weeks after a second positive serum β-hCG test
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 19 | 10
Participants | 0 | 2 | 5 | 7 | 0
Statistical Analysis 1: Comparison: Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled vs Placebo; Clinical pregnancy rates of the pooled LutrePulse 15 μg and 20 μg group were compared to placebo; Test type: Superiority — The hypotheses was tested using a stratified one-sided Fisher's exact test in the FAS including the randomization scheme as the stratification factor; p = 0.0383, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Biochemical Pregnancy Rate
Description: Proportion of subjects with a confirmed positive serum β-hCG test after luteinizing hormone (LH) surge.
Time Frame: Approximately 14 days after LH surge
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 19 | 10
Participants | 0 | 3 | 5 | 8 | 0
Statistical Analysis 1: Comparison: Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled vs Placebo; Biochemical pregnancy rates of the pooled LutrePulse 15 μg and 20 μg group were compared to placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0246, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: LH Surge Detection
Description: Proportion of subjects with a positive detection of LH surge, based on a Clearblue test which began when follicles with a mean diameter ≥14 mm were documented on TVUS.
Time Frame: Daily from Day 11 until first positive LH surge or until Day 39
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- LutrePulse 15 µg/Pulse: Gonadorelin acetate SC 15 µg/pulse as fixed dose, administered via. OmniPod pump
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 19 | 10
Participants | 3 | 7 | 6 | 13 | 0
Statistical Analysis 1: Comparison: Lutrepulse 15 μg/Pulse and 20 μg/Pulse Pooled vs Placebo; LH surge detection of the pooled LutrePulse 15 μg and 20 μg group were compared to placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0011, Fisher Exact — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Ovarian Follicular Development: Number of Follicles With a Mean Diameter Greater Than or Equal to (≥)14 mm
Description: Number of follicles with a mean diameter ≥14 mm collected from Days 10 or 11, until LH surge or Day 21.
Time Frame: From treatment Day 10 to treatment Day 21
Population: as for outcome 1
Measure: Median (Full Range); unit: follicles
Groups:
- Placebo: Placebo (SC 10, 15, or 20 μg/pulse as a fixed dose, administered via. OmniPod pump
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 10
follicles
  Day 10 | 0.0 [0 to 2] | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 0]
  Day 12: number analyzed (Participants) | 6 | 6 | 10 | 7
  Day 12 | 0.0 [0 to 1] | 0.5 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 0]
  Day 15: number analyzed (Participants) | 9 | 8 | 8 | 9
  Day 15 | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 0]
  Day 18: number analyzed (Participants) | 8 | 6 | 6 | 9
  Day 18 | 0.0 [0 to 1] | 1.0 [0 to 1] | 1.0 [0 to 2] | 0.0 [0 to 0]
  Day 21: number analyzed (Participants) | 4 | 6 | 3 | 7
  Day 21 | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 1] | 0.0 [0 to 0]
Statistical Analysis 1: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Day 10: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 10 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.1344, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 2: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Day 10: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 15 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.2726, Wilcoxon rank sum test — The p-value was based on the Wilcoxon rank sum test without stratification; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 3: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Day 10: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 20 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.3173, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 4: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Day 12: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 10 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.1275, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 5: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Day 12: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 15 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.1088, Wilcoxon rank sum test — The p-value was based on the Wilcoxon rank sum test without stratification; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 6: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Day 12: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 20 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.2374, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 7: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Day 15: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 10 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.0796, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 8: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Day 15: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 15 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.1757, Wilcoxon rank sum test — The p-value was based on the Wilcoxon rank sum test without stratification; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 9: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Day 15: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 20 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.0584, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 10: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Day 18: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 10 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.3711, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 11: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Day 18: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 15 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.0143, Wilcoxon rank sum test — The p-value was based on the Wilcoxon rank sum test without stratification; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 12: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Day 18: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 20 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.0060, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 13: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Day 21: Number of follicles with a mean diameter ≥14 mm in the LutrePulse 20 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.1573, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test

7. Secondary Outcome: Ovarian Follicular Development: Number of Dominant Follicles With a Mean Diameter of ≥18 mm
Description: Number of dominant follicles with a mean diameter ≥18 mm collected from Days 10 or 11, until LH surge or Day 21.
Time Frame: From treatment Day 10 to treatment Day 21
Population: as for outcome 1
Measure: Median (Full Range); unit: follicles
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 10
follicles
  Day 10 | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 0] | 0.0 [0 to 0]
  Day 12: number analyzed (Participants) | 6 | 6 | 10 | 7
  Day 12 | 0.0 [0 to 0] | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 0]
  Day 15: number analyzed (Participants) | 9 | 8 | 8 | 9
  Day 15 | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 0]
  Day 18: number analyzed (Participants) | 8 | 6 | 6 | 9
  Day 18 | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 0]
  Day 21: number analyzed (Participants) | 4 | 6 | 3 | 7
  Day 21 | 0.0 [0 to 1] | 0.0 [0 to 1] | 0.0 [0 to 0] | 0.0 [0 to 0]
Statistical Analysis 1: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Day 12: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 15 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.4142, Wilcoxon rank sum test — The p-value was based on the Wilcoxon rank sum test without stratification; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 2: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Number of follicles with a mean diameter ≥18 mm in the LutrePulse 20 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.2374, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 3: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Day 15: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 10 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.2636, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 4: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Day 15: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 15 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.4795, Wilcoxon rank sum test — The p-value was based on the Wilcoxon rank sum test without stratification; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 5: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Day 15: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 20 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.3173, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 6: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Day 18: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 10 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.3711, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 7: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Day 18: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 15 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.4142, Wilcoxon rank sum test — The p-value was based on the Wilcoxon rank sum test without stratification; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 8: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Day 18: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 20 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.0838, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 9: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Day 21: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 10 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.3173, Wilcoxon rank sum test — The p-value was based on the stratified (by randomization scheme) Wilcoxon rank sum test; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test
Statistical Analysis 10: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Day 21: Number of follicles with a mean diameter ≥18 mm in the LutrePulse 15 μg group was compared to placebo, using Wilcoxon's rank sum test; Test type: Superiority; p = 0.3778, Wilcoxon rank sum test — The p-value was based on the Wilcoxon rank sum test without stratification; SAS PROC FREQ with modified ridit score (MODRIDIT option) was used for the stratified Wilcoxon rank sum test

8. Secondary Outcome: Luteal Phase Support: Maximum P4 Levels
Description: Maximum of post-dose P4 levels collected on treatment Days 19 to 27 are presented.
Time Frame: Treatment Days 19, 21, 23, 25, and 27
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Groups:
- LutrePulse 10 µg/Pulse: Gonadorelin acetate SC 10 µg/pulse as a fixed dose, administered via. OmniPod
- LutrePulse 15 µg/Pulse: Gonadorelin acetate SC 15 µg/pulse as a fixed dose, administered via. OmniPod
- LutrePulse 20 µg/Pulse: Gonadorelin acetate SC 20 µg/pulse as a fixed dose, administered via. OmniPod
- Placebo: Placebo (SC 10, 15, or 20 μg/pulse as a fixed dose, administered via. OmniPod)
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 10
ng/mL | 0.40 [0.1 to 12.9] | 2.40 [0.4 to 18.5] | 8.00 [0.1 to 21.7] | 0.30 [0.1 to 0.4]
Statistical Analysis 1: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Maximum P4 levels in the LutrePulse 10 µg group were compared to placebo using an analysis of covariance (ANCOVA) model including the randomization scheme and treatment group as factors and baseline value as covariate; Test type: Superiority; p = 0.6732, ANCOVA — p-value for the LutrePulse 10 µg group compared to placebo based on the fitted linear model were reported; PROC GLM was used for ANCOVA; Least square mean (LSM) difference = 1.35, 95% CI 2-sided [-5.16 to 7.87] — The LSM difference on the treatment groups and 95% confidence interval (CI) for the LutrePulse 10 µg group compared to placebo based on the fitted linear model were reported. Type III sum-of-squares for the LSMs were used for statistical comparisons
Statistical Analysis 2: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Maximum P4 levels in the LutrePulse 15 µg group were compared to placebo using an ANCOVA model including treatment group as factors and baseline value as covariate; Test type: Superiority; p = 0.0814, ANCOVA — p-value for the LutrePulse 15 µg group compared to placebo based on the fitted linear model were reported; PROC GLM was used for ANCOVA; LSM = 5.70, 95% CI 2-sided [-0.76 to 12.15] — The LSM difference on the treatment groups and 95% CI for the LutrePulse 15 µg group compared to placebo based on the fitted linear model were reported. Type III sum-of-squares for the LSMs were used for statistical comparisons
Statistical Analysis 3: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Maximum P4 levels in the LutrePulse 20 µg group were compared to placebo using an ANCOVA model including the randomization scheme and treatment group as factors and baseline value as covariate; Test type: Superiority; p = 0.0223, ANCOVA — p-value for the LutrePulse 20 µg group compared to placebo based on the fitted linear model were reported; PROC GLM was used for ANCOVA; LSM difference = 7.55, 95% CI 2-sided [1.16 to 13.93] — The LSM difference on the treatment groups and 95% CI for the LutrePulse 20 µg group compared to placebo based on the fitted linear model were reported. Type III sum-of-squares for the LSMs were used for statistical comparisons

9. Secondary Outcome: Luteal Phase Support: Mean P4 Levels
Description: Mean of post-dose P4 levels collected on treatment Days 19 to 27 are presented.
Time Frame: Median post-dose P4 values across Treatment Days 19, 21, 23, 25, and 27
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Groups:
- LutrePulse 20 µg/Pulse: Gonadorelin acetate SC 20 µg/pulse as a fixed dose, , administered via. OmniPod
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 10
ng/mL | 0.313 [0.10 to 8.06] | 1.440 [0.26 to 8.50] | 3.920 [0.10 to 14.80] | 0.233 [0.10 to 0.40]
Statistical Analysis 1: Comparison: LutrePulse 10 µg/Pulse vs Placebo; Mean P4 levels in the LutrePulse 10 µg group were compared to placebo using an ANCOVA model including the randomization scheme and treatment group as factors and baseline value as covariate; Test type: Superiority; p = 0.7355, ANCOVA — p-value for the LutrePulse 10 µg group compared to placebo based on the fitted linear model were reported; PROC GLM was used for ANCOVA; LSM difference = 0.679, 95% CI 2-sided [-3.404 to 4.762] — The LSM difference on the treatment groups and 95% CI for the LutrePulse 10 µg group compared to placebo based on the fitted linear model were reported. Type III sum-of-squares for the LSMs were used for statistical comparisons
Statistical Analysis 2: Comparison: LutrePulse 15 µg/Pulse vs Placebo; Mean P4 levels in the LutrePulse 15 µg group were compared to placebo using an ANCOVA model including treatment group as factors and baseline value as covariate; Test type: Superiority; p = 0.1980, ANCOVA — p-value for the LutrePulse 15 µg group compared to placebo based on the fitted linear model were reported; PROC GLM was used for ANCOVA; LSM difference = 2.602, 95% CI 2-sided [-1.444 to 6.648] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: LutrePulse 20 µg/Pulse vs Placebo; Mean P4 levels in the LutrePulse 20 µg group were compared to placebo using an ANCOVA model including the randomization scheme and treatment group as factors and baseline value as covariate; Test type: Superiority; p = 0.0187, ANCOVA — p-value for the LutrePulse 10 µg group compared to placebo based on the fitted linear model were reported; PROC GLM was used for ANCOVA; LSM difference = 4.880, 95% CI 2-sided [0.878 to 8.882] — [estimate comment as in outcome 8, analysis 3]

10. Secondary Outcome: Change From Baseline in Follicle-stimulating Hormone (FSH)
Description: FSH change from baseline in relation to the first dose (pulse) on Day 1 and Day 10
Time Frame: Baseline (pre-dose), Treatment Day 1, Treatment Day 10
Population: as for outcome 1
Measure: Median (Full Range); unit: IU/L
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 10
IU/L
  FSH (Day 1) | 1.30 [0.0 to 7.7] | 5.40 [0.0 to 9.9] | 2.70 [0.0 to 5.7] | 0.10 [0.0 to 0.6]
  FSH (Day 10) | 0.04 [-0.8 to 0.8] | -0.04 [-0.3 to 0.4] | 0.04 [-0.7 to 0.6] | -0.01 [-0.1 to 0.1]
Statistical Analysis 1: Comparison: LutrePulse 10 µg/Pulse vs Placebo; The mean change in FSH levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 10 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.8772, ANCOVA — The p-value was derived from an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; LSM difference = 0.03, 95% CI 2-sided [-0.39 to 0.46] — LSM difference and CIs were derived from an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate
Statistical Analysis 2: Comparison: LutrePulse 15 µg/Pulse vs Placebo; The mean change in FSH levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 15 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.7805, ANCOVA — [p-value comment as in outcome 10, analysis 1]; LSM difference = 0.07, 95% CI 2-sided [-0.44 to 0.58] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: LutrePulse 20 µg/Pulse vs Placebo; The mean change in FSH levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 20 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.6095, ANCOVA — [p-value comment as in outcome 10, analysis 1]; LSM difference = 0.12, 95% CI 2-sided [-0.35 to 0.58] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Change From Baseline in LH
Description: LH change from baseline in relation to first dose (pulse) on Day 1 and Day 10
Time Frame: Baseline (pre-dose), Treatment Day 1, Treatment Day 10
Population: as for outcome 1
Measure: Median (Full Range); unit: IU/L
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 10
IU/L
  Day 1 | 1.85 [0.2 to 22.6] | 7.90 [0.4 to 23.6] | 5.15 [0.6 to 12.4] | 0.05 [-0.2 to 0.3]
  Day 10 | 0.00 [-2.9 to 1.6] | 0.58 [-1.7 to 1.9] | 0.03 [-0.9 to 1.7] | 0.00 [-1.0 to 0.0]
Statistical Analysis 1: Comparison: LutrePulse 10 µg/Pulse vs Placebo; The mean change in LH levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 10 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.1520, ANCOVA — [p-value comment as in outcome 10, analysis 1]; LSM difference = 0.51, 95% CI 2-sided [-0.20 to 1.22] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: LutrePulse 15 µg/Pulse vs Placebo; The mean change in LH levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 15 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.0221, ANCOVA — [p-value comment as in outcome 10, analysis 1]; LSM difference = 0.93, 95% CI 2-sided [0.14 to 1.72] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: LutrePulse 20 µg/Pulse vs Placebo; The mean change in LH levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 20 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.0316, ANCOVA — [p-value comment as in outcome 10, analysis 1]; LSM difference = 0.76, 95% CI 2-sided [0.07 to 1.44] — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Mean Serum FSH and LH Levels
Description: Mean FSH and LH levels on Day 1 and Day 10.
Time Frame: Treatment Days 1 and Day 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 10
IU/L
  FSH (Baseline) | 1.59 (1.793) | 1.47 (1.112) | 2.48 (2.235) | 1.35 (1.520)
  FSH (Day 1) | 3.64 (4.010) | 6.20 (3.929) | 5.38 (2.565) | 1.52 (1.673)
  FSH (Day 10): number analyzed (Participants) | 9 | 9 | 10 | 9
  FSH (Day 10) | 4.00 (1.495) | 5.07 (2.530) | 5.24 (1.124) | 1.67 (1.796)
  LH (Baseline) | 0.54 (0.669) | 0.27 (0.179) | 0.93 (0.954) | 0.73 (1.063)
  LH (Day 1) | 6.27 (9.507) | 8.82 (7.348) | 6.12 (3.745) | 0.79 (1.026)
  LH (Day 10): number analyzed (Participants) | 9 | 9 | 10 | 9
  LH (Day 10) | 4.12 (3.931) | 4.69 (2.692) | 4.07 (2.335) | 0.82 (1.037)

13. Secondary Outcome: Estradiol (E2) Serum Levels
Description: E2 serum levels on Day 1 and Day 10.
Time Frame: At treatment Day 1 and Day 10
Population: as for outcome 1
Measure: Median (Full Range); unit: pmol/L
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 10
pmol/L
  Day 1 (pre-dose) | 36.50 [36.5 to 169.0] | 88.00 [36.5 to 147.0] | 81.00 [36.5 to 92.0] | 122.50 [36.5 to 198.0]
  Day 10 (pre-dose) | 106.00 [36.5 to 697.0] | 202.00 [84.0 to 499.0] | 136.00 [36.5 to 323.0] | 128.00 [36.5 to 224.0]
Statistical Analysis 1: Comparison: LutrePulse 10 µg/Pulse vs Placebo; The mean change in E2 levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 10 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.3147, ANCOVA — [p-value comment as in outcome 10, analysis 1]; LSM difference = 73.00, 95% CI 2-sided [-72.66 to 218.65] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: LutrePulse 15 µg/Pulse vs Placebo; The mean change in E2 levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 15 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.2290, ANCOVA — [p-value comment as in outcome 10, analysis 1]; LSM difference = 95.18, 95% CI 2-sided [-63.01 to 253.36] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: LutrePulse 20 µg/Pulse vs Placebo; The mean change in E2 levels from Day 10 pre-treatment (prior to first dose) in the LutrePulse 20 μg/Pulse group was compared to placebo using an ANCOVA model with randomization scheme and treatment as factors and baseline value as covariate; Test type: Superiority; p = 0.5066, ANCOVA — [p-value comment as in outcome 10, analysis 1]; LSM difference = 46.99, 95% CI 2-sided [-95.64 to 189.61] — [estimate comment as in outcome 10, analysis 1]

14. Secondary Outcome: Type, Intensity, and Frequency of Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a subject taking part in a clinical trial. Proportion of subjects with any AE (serious or non-serious) and intensity of AEs (classified as mild, moderate or severe) are presented.
Time Frame: From treatment Day 1 to end-of-trial, approximately 10 weeks
Population: The safety analysis set comprised all randomized subjects who received at least one pulsatile delivery of IMP. The number count is based on the actual treatment subjects received: one subject randomized to LutrePulse 15 µg/Pulse had received placebo and was moved to the placebo group in the safety analysis set (LutrePulse 15 µg/Pulse: n=8, Placebo: n=11)
Measure: Count of Participants; unit: Participants
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 10 | 8 | 10 | 11
Participants
  Any AE | 5 | 3 | 4 | 4
  Non-serious AE | 5 | 3 | 4 | 4
  Serious AE | 0 | 0 | 0 | 0
  Intensity (Mild) | 5 | 1 | 2 | 1
  Intensity (Moderate) | 0 | 2 | 2 | 2
  Intensity (Severe) | 0 | 0 | 0 | 1

15. Secondary Outcome: Hematology, Clinical Chemistry, and Urinalysis
Description: Proportion of subjects with markedly abnormal changes in hematology, clinical chemistry, and urinalysis.
Time Frame: From treatment Day 1 to end-of-trial, approximately 10 weeks
Population: as for outcome 14
Measure: Number; unit: participants
Groups:
- LutrePulse 10 µg/Pulse: Gonadorelin acetate SC 10 µg/pulse as fixed dose, administered via. OmniPod pump
- LutrePulse 20 µg/Pulse: Gonadorelin acetate SC 20 µg/pulse as fixed dose, administered via. OmniPod pump
- Placebo: Placebo (SC 10, 15, or 20 μg/pulse as a fixed dose, , administered via. OmniPod pump)
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 10 | 8 | 10 | 11
participants
  Hematology: number analyzed (Participants) | 9 | 8 | 10 | 11
  Hematology | 0 | 0 | 0 | 0
  Serum chemistry (Sodium, <=130 mmol/L): number analyzed (Participants) | 10 | 7 | 10 | 10
  Serum chemistry (Sodium, <=130 mmol/L) | 0 | 1 | 0 | 0
  Urinalysis (Protein,mg/dL, -ve to +ve [post-dose]): number analyzed (Participants) | 10 | 8 | 9 | 10
  Urinalysis (Protein,mg/dL, -ve to +ve [post-dose]) | 2 | 0 | 1 | 0
  Urinalysis (Specific Gravity <=1.005): number analyzed (Participants) | 9 | 8 | 10 | 11
  Urinalysis (Specific Gravity <=1.005) | 0 | 1 | 1 | 0

16. Secondary Outcome: Frequency and Severity of Ovarian Hyperstimulation Syndrome (OHSS)
Description: Proportion of subjects reporting OHSS classified as mild, moderate, or severe.
Time Frame: From treatment Day 1 to end-of-trial, approximately 10 weeks
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
Number analyzed (Participants) | 10 | 8 | 10 | 11
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) occurred after the start of IMP administration and within 5 days after the last dose, or a pre-treatment AE or pre-existing medical conditioning the worsened in intensity after the start of IMP and within 5 days after the last dose
Description: TEAEs were defined as AEs that occurred after the start of IMP administration and within 5 days after the last dose.
  All subjects who received at least one pulsatile injection delivery of IMP were included in safety analysis set and were analyzed according to the actual treatment received. One subject randomized to LutrePulse 15 µg/Pulse had received placebo and was moved to the placebo group in the safety analysis set (LutrePulse 15 µg/Pulse: n=8, Placebo: n=11).
Arm/Group | LutrePulse 10 µg/Pulse | LutrePulse 15 µg/Pulse | LutrePulse 20 µg/Pulse | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/8 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 5/10 | 3/8 | 4/10 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LutrePulse 10 µg/Pulse (N=10) | LutrePulse 15 µg/Pulse (N=8) | LutrePulse 20 µg/Pulse (N=10) | Placebo (N=11)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distesion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Adnexa uteri pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flushes (Vascular disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.

DOCUMENTS (2):
  • Study Protocol (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT01976728/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT01976728/SAP_001.pdf